CLINICAL TRIAL: NCT05811416
Title: Observational, Multicenter Study to Describe the Persistence in Relapsing Remitting Multiple Sclerosis Naive Patients With Low-moderate Activity Treated With Ozanimod (Zeposia®) in Clinical Practice in Spain
Brief Title: A Study to Describe the Persistence With Ozanimod Treatment in Relapsing-Remitting Multiple Sclerosis (RRMS) Participants
Acronym: AppreZiate
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-066
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
Keywords: Ozanimod; Zeposia; Relapsing-remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort 1: Participants that have initiated ozanimod.

SUMMARY:
The purpose of the study is to collect clinical data on the persistence with ozanimod treatment, as well as to describe its effects on participant-relevant outcome parameters in treatment-naïve participants with RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis (RRMS) diagnosis by 2017 revised McDonald criteria at the treatment start

  * Participant who started treatment with ozanimod for the first time 3 months (+/- 2 weeks) before inclusion, according to European Union (EU) Summary of Product Characteristics (SmPC) and/or Spanish therapeutic positioning report (TPR) recommendation and following routine clinical practice of the participating hospital
  * Low-to-moderate activity, defined as less than 2 relapses in the previous year before starting the treatment with ozanimod

Exclusion Criteria:

* Prior exposure to ozanimod or any other disease modifier treatment (DMT) for RRMS before starting treatment with ozanimod subject of this study
* Participant who has started ozanimod within a clinical trial

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates will be adult treatment-naïve participants diagnosed with RRMS who attend to a regular follow up visit at a Spanish participating hospital and who started treatment with ozanimod for the first time 3 months (+/- 2 weeks) before inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-11-09 (Estimated); Study Completion 2026-11-09 (Estimated)

PRIMARY OUTCOMES:
Time from ozanimod treatment initiation to ozanimod treatment permanent discontinuation | Up to 24 months
Percentage of participants on treatment with ozanimod at 24 months | At month 24

SECONDARY OUTCOMES:
Percentage of participants with ozanimod treatment at 3 and 12 months | At month 3 and month 12
Percentage of participants with ozanimod treatment discontinuation | Up to 24 months
Percentage of participants switching to treatment alternative | Up to 24 months
Annualized relapse rate at month 12 month and month 24 | At month 12 and month 24
Proportion of participants with an increase in Symbol Digit Modalities Test (SDMT) score of ≥4 points | At month 3, 12 and 24
Proportion of participants with a decrease SDMT score of ≥4 points | At month 3, 12 and 24
Proportion of participants with a stable SDMT score | At month 3, 12 and 24
Change from baseline in SDMT score at month 3, 12 and 24 | Baseline, Month 3, 12 and 24
Change from baseline in Neurofilament light (NfL) levels at month 6, 12 and 24 | Baseline, Month 6, 12 and 24
Proportion of participants with change of ≥1.0 point from baseline in expanded disability status scale (EDSS) score at Month 3, 12 and 24 | Baseline, Month 3, 12 and 24
Change from baseline in EDSS score at Month 3, 12 and 24 | Baseline, Month 3, 12 and 24
Change from baseline in number of new or enlarging hypointense T1 lesions at month 12 and 24 | Baseline, Month 12 and 24
Change from baseline in number of new or enlarging hypointense T2 lesions at month 12 and 24 | Baseline, Month 12 and 24
Change from baseline in number of new or enlarging gadolinium enhancing brain lesions at month 12 and 24 | Baseline, Month 12 and 24
Number of Participants with at least one Adverse Event (AE) | Up to 24 months
Number of Participants with AE that imply discontinuation of ozanimod | Up to 24 months
Description of sociodemographic characteristics of participants | Baseline, up to 24 months
Description of clinical characteristics of participants | Baseline, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Barcelona, Spain

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm